CLINICAL TRIAL: NCT02556528
Title: A Study to Assess the Feasibility of Using Health Coaching Sessions in Cancer Patients
Brief Title: Feasibility of Health Coaching in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PID: 11437
Record Dates: First submitted 2015-09-17; First posted 2015-09-22 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health Coaching (Experimental)
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Health Coaching

SUMMARY:
This is a study to assess the feasibility of using health coaching sessions in cancer patients. The investigators are investigating whether health coaching sessions can be delivered to this group of participants in a semi structured way. The investigators hope that the study will allow us to see whether such sessions can be delivered in a timely manner that is acceptable to patients and staff. The longer term aim for this work, should it prove feasible, is to conduct a randomised controlled trial to assess health coaching.

The participants for the study will be selected using purposive sampling. The investigators will select a sample of 10 patients. The participants will be patients at the Oxford University Hospitals NHS Trust who are prescribed oral anticancer therapy. The sample will include male and female patients and try to cover a range of ages from 18 upwards. It will cover patients taking a range of oral anticancer agents, for a range of different cancer indications. The sample will look at patients who are newly prescribed oral anticancer therapy through to patients who have been taking therapy for years.

Participants will be identified for the study by multidisciplinary staff members who are running oral education sessions or by non-medical prescribers who are seeing patients in clinic. These members of the multidisciplinary team (MDT) will be given lists of the types of participants the investigators are looking for in the study and where appropriate offer patients the opportunity to take part. Patients will be contacted prior to the end of their subsequent cycle of treatment about whether they wish to participate. Patients wishing to take part will be consented at their next clinic visit.

All participants will attend for their usual clinic visits throughout the study. Participants will additionally be offered up to 3 health coaching sessions for a maximum of three cycles or until treatment with their oral anticancer agent ends, whichever comes first.

At the end of study visit participants will be asked to attend a qualitative based interview to discuss the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to comply with the protocol for the duration of the study.
* Patient is willing and able to give written (signed and dated) informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with cancer.
* Patient prescribed an oral anticancer agent.

Exclusion Criteria:

* Patients who are unable to complete 1 cycle of oral anticancer therapy from the time of being approached about the trial.
* Patients who would be unable to participate in a health coaching session with a health coach for any reasons, including, difficulty understanding or speaking English, other communication difficulties or hearing problems.
* Other psychological, social or medical condition, that the Investigator considers would make the patient a poor trial candidate, could interfere with protocol compliance, could affect the patient's ability to give informed consent or may affect the interpretation of trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of health coaching intervention in cancer patients within the NHS | up to 4months (depending on length of each cycle of treatment). Patients will be seen at up to 4 consecutive clinic visits.
  To assess whether a 10 minute semi standardised health coaching session can be conducted with NHS cancer patients by pharmacists trained in health coaching and to gather the opinions of the patients and the health coaches as to whether the intervention is of benefit and warrants further investigation.
  Measures of feasibility include: Recruitment figures, logistics of conducting health coaching sessions, review of the recorded coaching sessions, attendance rates, qualitative analysis of reflection notes and end of study interview with patients, Patient activation measure at baseline and end of study.